CLINICAL TRIAL: NCT01196650
Title: A Double Blind, Polysomnographic, Three-Way Crossover Study to Compare the Efficacy of IN 10 003 to Placebo in Subjects With Insomnia Suffering From Difficulty in Falling Asleep and Staying Asleep
Brief Title: Comparison of IN 10 003 to Placebo in Subjects With Insomnia Suffering From Difficulty in Falling Asleep and Staying Asleep
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intec Pharma Ltd. (Industry)
Responsible Party: Hadas Friedman, Intec Pharma Ltd.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IN 10 003
Record Dates: First submitted 2010-09-05; First posted 2010-09-08 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2010-09

CONDITIONS: Subjects With Insomnia Suffering From Difficulty in Falling Asleep and Staying Asleep

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- 1 (Active Comparator): IN 10 003 formulation A
  Interventions: Drug: IN 10 003 formulation A
- 2 (Active Comparator): IN 10 003 formulation B
  Interventions: Drug: IN 10 003 formulation B
- 3 (Placebo Comparator): Placebo capsules
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: IN 10 003 formulation A
  Arms: 1
Drug: IN 10 003 formulation B
  Arms: 2
Drug: Placebo capsules
  Arms: 3

SUMMARY:
This study aims to assess the efficacy of IN 10 003 in improving sleep parameters in patients with Insomnia exhibiting both difficulty in falling asleep and staying asleep. The study will compare 2 formulations of the IN 10 003 to placebo

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 18 and 65 years of age
* Subjects that meet DSM IV diagnostic criteria for Insomnia
* Subjects that report a time in bed NLT 6.5 and NMT 9 hours
* Subjects that report on a one week sleep diary (on at least 3 of 7 nights) TST NMT 6.5 hours
* Subjects that report on a one week sleep diary (on at least 3 of 7 nights) Wake time after sleep >1.0 hour
* Subjects that report on a one week sleep diary (on at least 3 of 7 nights) NLT 30 minutes time to sleep onset
* On two nights of PSG screening a mean WASO of ≥60 minutes with neither night less than 45 minutes
* On two nights of PSG screening a mean LPS of ≥20 minutes with neither night less than 15 minutes
* On two nights of PSG screening a TST of NMT 6.5 hours on each of the two nights

Exclusion Criteria:

* Subject has a circadian rhythm disorder including shift work or the need to travel NLT 3 time zones during the course of the study
* Use of any drug known to effect sleep or wake functions within 5 half lives of the drug or two weeks, whichever comes first.
* Subject with a history (past year) of alcohol or substance abuse
* Subject that needs to smoke during the sleep period time
* Subject that reports habitual napping (more than 3 times per week)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-09

PRIMARY OUTCOMES:
Wake after sleep onset
  To determine the effect of IN 10 003 on Wake time After Sleep Onset (WASO) as the change from baseline for the mean of night 1 and 2 relative to placebo

SECONDARY OUTCOMES:
Objective and Subjective sleep parameters
  Total Sleep Time, Latency to Persistent Sleep, Absence of residual effects,

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Soroka University Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Assuta Medical Center, Tel Aviv